CLINICAL TRIAL: NCT07238881
Title: A Prospective, Randomized, Two-Cohort, Exploratory Clinical Study of Dalpiciclib Combined With Camrelizumab in Patients With Unresectable Hepatocellular Carcinoma Previously Treated With Immune Checkpoint Inhibitors
Brief Title: Dalpiciclib Plus Camrelizumab for HCC Patients Who Have Previously Received ICI Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-II -029
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellulcar Carcinoma
Keywords: Dalpiciclib; Camrelizumab; second-line treatment
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dalpiciclib +Camrelizumab (Experimental): Dalpiciclib 125mg, qd+Camrelizumab 200mg q2w
  Interventions: Drug: Dalpiciclib Isetionate Tablets; Drug: Camrelizumab (anti-PD-1 inhibitor)
- Low-Dalpiciclib +Camrelizumab (Experimental): Dalpiciclib 100mg, qd+Camrelizumab 200mg q2w
  Interventions: Drug: Dalpiciclib Isetionate Tablets; Drug: Camrelizumab (anti-PD-1 inhibitor)

INTERVENTIONS:
Drug: Dalpiciclib Isetionate Tablets — Dalpiciclib 125mg
  Arms: High-Dalpiciclib +Camrelizumab
Drug: Dalpiciclib Isetionate Tablets — Dalpiciclib 100mg
  Arms: Low-Dalpiciclib +Camrelizumab
Drug: Camrelizumab (anti-PD-1 inhibitor) — Camrelizumab 200mg

SUMMARY:
While immune-based therapies (including targeted-immune or dual-immune regimens) have become first-line standard for advanced hepatocellular carcinoma (HCC), there is a lack of high-level evidence to guide second-line treatment after progression on immune checkpoint inhibitors (ICIs).

Preclinical studies suggest synergistic antitumor activity between CDK4/6 inhibitors and PD-1/PD-L1 blockade. However, no clinical studies have yet evaluated the combination of dalpiciclib and camrelizumab in this setting.

To address this unmet need and explore novel second-line strategies for advanced HCC, we plan to conduct an exploratory clinical trial investigating the efficacy and safety of dalpiciclib plus camrelizumab in patients with unresectable HCC previously treated with ICIs.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Patients who have previously received first-line treatment with ICI treatments (including PD-1/PD-L1/CTLA-4) and who have shown tumor progression as confirmed by imaging studies.
* Eastern Cooperative Oncology Group performance status of 0 to 1
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS is the length of time from the date of randomization until death from any cause.
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
Adverse events | 30 days
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China